CLINICAL TRIAL: NCT04297020
Title: Brain Health in Breast Cancer Survivors: Interaction of Menopause and Endocrine Therapy
Brief Title: Brain Health in Breast Cancer Survivors
Status: Recruiting | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-001004; K08CA241337 (NIH); NCI-2020-01501 (Registry Identifier: CTRP)
Record Dates: First submitted 2020-02-28; First posted 2020-03-05 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Impairment; Cognitive Function
Keywords: Breast cancer; endocrine therapy
MeSH Terms: conditions — Cognitive Dysfunction; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Pre-menopausal BCS + ET: Pre-menopausal Breast Cancer Survivor (BCS) who have undergone Endocrine Therapy (ET)
- Post-menopausal BCS + ET: Post-menopausal Breast Cancer Survivor (BCS) who have undergone Endocrine Therapy (ET)
- Pre-menopausal Healthy Control: Pre-menopausal healthy control group
- Post-menopausal Healthy Control: Post-menopausal healthy control group

SUMMARY:
Endocrine therapy (ET) is widely used to treat hormone receptor positive breast cancer and prevent recurrence by downregulating estrogen function. However, ETs readily cross the blood brain barrier and interfere with the action of estrogen in the brain. Estrogen supports cognition and menopausal status is closely linked to cognitive health in women. This has raised concern that anti-estrogen ETs may affect cognition and brain health in breast cancer survivors. However, evidence across existing studies is inconsistent and these effects remain poorly understood. The incomplete understanding of the effects of ET are likely due to limitations of earlier studies - namely, the under-appreciation of the role of menopausal status and insensitivity of standard cognitive measures. This research project will address these earlier limitations by specifically comparing ET effects by menopausal status, and using highly sensitive, task-related functional magnetic resonance imaging (fMRI) measures to assess the effects of ET on brain function.

DETAILED DESCRIPTION:
Endocrine therapy (ET) is widely used to treat hormone receptor positive breast cancer and prevent recurrence by downregulating estrogen function. However, ETs readily cross the blood brain barrier and interfere with the action of estrogen in the brain. Estrogen supports cognition and menopausal status is closely linked to cognitive health in women. This has raised concern that anti-estrogen ETs may affect cognition and brain health in breast cancer survivors. However, evidence across existing studies is inconsistent and these effects remain poorly understood. The incomplete understanding of the effects of ET are likely due to limitations of earlier studies - namely, the under-appreciation of the role of menopausal status and insensitivity of standard cognitive measures. This research project will address these earlier limitations by specifically comparing ET effects by menopausal status, and using highly sensitive, task-related fMRI measures to assess the effects of ET on brain function.

This study is a cross-sectional study in a 2x2 factorial design comparing menopausal status (pre and post) and patient group (breast cancer survivors on ET and healthy controls matched on age, race, education, and time since final menstrual period (post only)). The investigators will use sensitive fMRI measures of brain activity during a working memory task - measures successfully used to reveal the effects of menopause and estrogen changes in healthy women, but yet to be extensively used to study the effects of ET.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-65
* Fluent in English
* Adequate vision/hearing to complete testing

Exclusion Criteria:

* History of major or mild neurocognitive disorder or dementia
* Diagnosis of major neurological condition (e.g., epilepsy, Parkinson's Disease, stroke)
* Diagnosis of a major psychiatric disorder (e.g., bipolar disorder, schizophrenia)
* Untreated/unstable unipolar depression or anxiety
* Prior history of cancer or chemotherapy (for controls, any history)
* History of a learning disorder
* History of head injury with loss of consciousness >20 minutes
* History of salpingo-oophorectomy or hysterectomy
* A cardiac pacemaker
* Implanted electronic device
* Claustrophobia
* Currently pregnant
* Orbital metal implant or other metallic foreign bodies

Additional exclusion criteria for controls: current use of a contraceptive agent that interferes with endogenous hormonal fluctuation (e.g., oral contraceptive pill) or precludes determination of menstrual pattern (e.g., hormonally secreting intrauterine device), or current treatment with systemic estrogen replacement therapy.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pre-menopausal and post-menopausal breast cancer survivors who are undergoing endocrine therapy.
Study Population: Pre-menopausal and post-menopausal breast cancer survivors who are undergoing endocrine therapy will be compared to healthy control group matched by age, race, education and time since final menstrual period (post only).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Brain activity comparison between breast cancer survivors undergoing endocrine therapy and healthy matched control subject. | Day 1
  To compare brain activity using fMRI during a working memory task between breast cancer survivors on ET and matched healthy controls, and examine the interaction of menopausal status.
Cognitive function comparison between breast cancer survivors undergoing endocrine therapy and healthy matched control subject. | Day 1
  To compare cognitive function between breast cancer survivors on ET and matched healthy controls, and examine the interaction of menopausal status.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Van Dyk, PhD, Principal Investigator — University of California at Los Angeles
Locations (1):
- University of California at Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No